CLINICAL TRIAL: NCT05622396
Title: A Pilot Feasibility Study of a Co-constructed Program (Patients - Experts) of Mindfulness Meditation Adapted to Patients With Parkinson's Disease.
Brief Title: Feasibility of an Adapted Mindfulness Program to Parkinson's Disease
Acronym: MAdaPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/54
Record Dates: First submitted 2022-10-27; First posted 2022-11-18 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Mindfulness; Adapted MBSR program; Feasibility; Efficacy
MeSH Terms: conditions — Parkinson Disease | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBSR program adapted (Experimental): 8 week program with weekly sessions of 2h30 and a full day of practice designed from the analysis of the post-program interviews
  Interventions: Procedure: Mindfulness Based Stress Reduction

INTERVENTIONS:
Procedure: Mindfulness Based Stress Reduction — Inspired by the standard Mindfulness Based Stress Reductio program, the study MAdaPARK is a 8 week program with weekly sessions of 2h30 and a full day of practice designed from the analysis of the post-program interviews carried out as part of the M-PARK study,as well as the reflections of the working group specially set up for this purpose. Several areas of adaptation have been identified: shorter mediations, a break time during the sessions, more times for exchanges, a more developed practice in movement, and finally, more important work based on self-esteem and self-compassion.

SUMMARY:
The objective of this study is to determine the feasibility (primary objective) and the effects (secondary objectives) of an Mindfulness Based Stress Reduction (MBSR) program adapted specifically for patients with Parkinson's disease.

DETAILED DESCRIPTION:
In Parkinson's disease (PD) the psychological distress (anxiety and depression), is particularly impacting and often resistant to conventional drug treatment explaining the growing interest of patients in non-drug methods, such as mindfulness meditation. The Mindfulness Based Stress Reduction (MBSR) program has been evaluated in Parkinson's disease, showing main effects on anxiety and depression symptoms. These data remain, however, still fragile, particularly in terms of methodological robustness and number of patients involved and variable size of effects. A clinical trial was recently conducted at the Bordeaux University Hospital with 28 patients with Parkinson's disease . Preliminary results suggest that a program tailored specifically to the expectations and needs of patients with Parkinson's disease could, optimize accessibility, acceptability, and patient compliance for this type of approach while preserving clinical efficacy on anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from Parkinson's disease,
* Patient aged over 18 and under 80,
* Patient with a Hoehn and Yahr Stage of 1 to 3,
* Patient affiliated or beneficiary of the social security system,
* Patient having signed a free, informed and written consent

Exclusion Criteria:

* Patient with severe motor fluctuations (i.e. scoring 4 to at least one of the following items of part IV of the Movement Disorder Society Unified Parkinson Disease Rating Scale: 4.1 and 4.2 for dyskinesias; 4.3, 4.4 and 4.5 for motor fluctuations),
* Patient with acute depression not stabilized by treatment or dating from less than 6 months,
* Patient with non-stabilized psycho-behavioral disorders (hallucinations, psychoses, impulse control disorders) dating from less than 6 months,
* Patient with major cognitive impairment (Montreal Cognitive Assessment ≤24),
* Patient who has already participated in a structured mindfulness meditation program
* Patient placed under judicial safeguard, guardianship or curator ship,
* Pregnant or breastfeeding women.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assess MBSR program | Month 4
  The rate of patients who have completed the entire MBSR program "adapted"

SECONDARY OUTCOMES:
Attendance rate | Month 3
  Number of days of practice and daily meditation time.
Program tolerance | month 1 at month 2
  Number of side effects and the difficulties
Relevance of the adaptations put in place | month 3
  It will be evaluated from the analysis of feelings and impressions of patients . These different elements will be obtained from the analysis of the semi-directed interviews (qualitative analysis).
Beck Depression Inventory | Day 0 and month 3
  Assessment depressive symptoms, minimum value 0 and maximum value 36
Parkinson Anxiety Scale (PAS) | Day 0 and month 3
  Assessment anxiety symptoms,minimum value 0 and maximum value 48
Parkinson's Disease Sleep Scale | Day 0 and month 3
  Assessment sleep, minimum value 0 and maximum value 60
Parkinson Disease Questionnaire | Day 0 and month 3
  Assessment quality of life, minimum value 0 and maximum value 156
Movement Disorder Society Unified Parkinson Disease Rating Scale | Day 0 and month 3
  Assessment motor and non-motor symptoms of Parkinson Disease
King's college Parkinson's disease Pain Scale | Day 0 and month 3
  Assessment pain, minimum value 0 and maximum value 168
Number of Anti-parkinsonian and psychotropic treatments | Day 0 and month 3

CONTACTS AND LOCATIONS:
Overall Officials: François TISON, Pr, Principal Investigator — Université Hospital, Bordeaux
Locations (1):
- Xavier Arnozan Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No